CLINICAL TRIAL: NCT05630404
Title: Efficacy of Surgical Injection Lumbar Erector Spinae Plane Block for Pain Management Following Lumbar Spinal Fusion Surgery
Brief Title: Efficacy of Surgical Injection Lumbar Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Mursel Ekinci, MD, Assoc Prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BursaCityHospital
Record Dates: First submitted 2022-11-01; First posted 2022-11-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Spine Instability; Lumbar Spinal Stenosis; Lumbar Spine Degeneration
Keywords: Lumbar spinal fusion surgery; Postoperative analgesia; Erector spina plan block
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: There are three models for this study. The first group is ultrasound guided erector spinae plane block group. The second one is surgical injection erector spinae plane block group. The third one is the no intervention control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, investigators and the pain nurse who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group IE= Surgical Injection ESPB (Active Comparator): Patients will be administered tenoxicam 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit.Tenoxicam 20 mg and a dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia.
  Interventions: Drug: Surgical ESPB
- Group UE= US guided ESPB (Active Comparator): Patients will be administered tenoxicam 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit.Tenoxicam 20 mg and a dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia.Tenoxicam 20 mg and a dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia.
  Interventions: Drug: US guided ESPB
- Group C = Control group (No Intervention): Tenoxicam 20 mg and a dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia.
  Patients will be administered tenoxicam 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit.

INTERVENTIONS:
Drug: Surgical ESPB — In group IE, transverse processes will be palpated before sewing the surgical incision by the surgery team. The local anesthetic solution will be administered after the needle contacts the transverse process and its location is confirmed by negative aspiration. Once the needle tip will be placed within the interfacial plane and after careful aspiration to rule out intravascular needle placement, 5 mL of solution will be injected the proper injection site. Local anesthetic solution will be injected at 4 levels along the surgical incision line. A dose of 0.25% bupivacaine 20 mL will be injected in each side (total 40 mL).
  Tenoxicam 20 mg and a dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia.
  Arms: Group IE= Surgical Injection ESPB
Drug: US guided ESPB — US guided ESP block will be performed. US probe will be placed longitudinally 2-3 cm lateral to the L3 transverse process. Erector spinae muscle will be visualized on the hyperechoic transverse process. The block needle will be inserted cranio caudal direction and then for correction of the needle 2 ml saline will be enjected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 20 ml %0.25 bupivacaine will be administered for block in each side (total 40 mL).
  Tenoxicam 20 mg and a dose of 100 mg tramadol intravenously will be performed to all patients 30 min before the end of the surgery for postoperative analgesia.
  Arms: Group UE= US guided ESPB

SUMMARY:
Lumbar spinal surgery is one of the operations performed for the treatment of leg and back pain. Severe pain may occur at postoperative period in patients following lumbar fusion surgery.

The ultrasound(US) guided erector spina plan block (ESPB) is injected with a local anesthetic into the deep fascia of the erector spinae. Visualization of sonoanatomy with US is simple and the spread of local anesthetic solution can be seen easily the deep fascia of the erector spinae. In the literature, it has been reported that ESPB provides effective analgesia after lumbar spine surgery. The surgical team visualizes the transverse processes and erector spina muscle during surgery.

The aim of this study is to compare US-guided ESPB and surgical infiltrative ESPB for postoperative analgesia management after lumbar spinal fusion surgery.

DETAILED DESCRIPTION:
Lumbar spinal surgery is one of the operations performed for the treatment of leg and back pain. Severe pain may occur at postoperative period in patients following lumbar fusion surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay, thus complications due to hospitalization such as infection and thromboembolism may be reduced.

Parenteral opioids are generally preferred in the management of acute postoperative pain. However opioids have undesired adverse events such as nausea, vomiting, itching, sedation and respiratory depression (opioid-related adverse events). Regional anesthesia techniques may be preferred as the use of ultrasound (US) increases in daily anesthesia practice.

The ultrasound(US) guided erector spina plan block (ESPB) is injected with a local anesthetic into the deep fascia of the erector spinae. Visualization of sonoanatomy with US is simple and the spread of local anesthetic solution can be seen easily the deep fascia of the erector spinae. In the literature, it has been reported that ESPB provides effective analgesia after lumbar spine surgery. The surgical team visualizes the transverse processes and erector spina muscle during surgery. The erector spina plane block can be performed by administering local anesthetic solution between the transverse process and the erector spina muscle.

The aim of this study is to compare US-guided ESPB and surgical infiltrative ESPB for postoperative analgesia management after lumbar spinal fusion surgery. The primary aim is to compare perioperative and postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* 2 or 3 levels of posterior lumbar spinal fusion surgery under general anesthesia

Exclusion Criteria:

* history of bleeding diathesis
* receiving anticoagulant treatment
* known local anesthetics and opioid allergy
* infection of the skin at the site of the needle puncture
* pregnancy or lactation
* patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | Change from Baseline Opioid Consumption for Postoperative 24 hours.
  Postoperative opioid consumption will be evaluated at postoperative 24 h period

SECONDARY OUTCOMES:
Visual analogue scores (VAS) | postoperative 1, 2, 4, 8, 16 and 24 hours
  VAS score (0 = no pain, 10 = the most severe pain felt)

CONTACTS AND LOCATIONS:
Locations (1):
- Mursel Ekinci, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigator's will not share IPD

REFERENCES:
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517
- [Background] Finnerty DT, Buggy DJ. Efficacy of the erector spinae plane (ESP) block for quality of recovery in posterior thoraco-lumbar spinal decompression surgery: study protocol for a randomised controlled trial. Trials. 2021 Feb 17;22(1):150. doi: 10.1186/s13063-021-05101-2. PMID 33596968